CLINICAL TRIAL: NCT03227627
Title: Outcomes of Using LNMES on Tracheostomized Children
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We decided to go to another direction.
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Sarah Stulberger, Co-Principal Investigator, Children's Hospital Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHLA-17-00081
Record Dates: First submitted 2017-02-27; First posted 2017-07-24 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Trachea
MeSH Terms: conditions — Tracheal Diseases

STUDY DESIGN:
Intervention Model Description: One group of children (Group A) will receive 24 sessions of NMES for combined with traditional therapy including oral motor exercises and laryngeal exercises will be performed to the participants. The other group (Group B) will be receiving 24 sessions of traditional dysphagia therapy. After the 24 sessions, participants will have a repeat MBSS and results will be scored using the Pen-Asp scale and FOIS scale. Both the control group and experimental group will answer the PSI-4 after the repeat MBSS.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- VitalStim (Experimental): One group of children (Group A) will receive 24 sessions of NMES for combined with traditional therapy including oral motor exercises and laryngeal exercises will be performed to the participants. The equipment to be used for NMES is VitalStim®. VitalStim is a product of Empi®. VitalStim® therapy involves the placement of electrodes to the muscles of the throat that is attached to a device that provides electrical stimulation. The intensity will be increased according to the subject's tolerance and when a "therapeutic" level is reached. Signs of reaching therapeutic level include changes in audible quality of swallows, triggers of swallows, and changes in quality of voice. This therapy is to be performed by a VitalStim® certified practitioner.
  Interventions: Device: VitalStim
- Traditional therapy (Active Comparator): The other group (Group B) will be receiving 24 sessions of traditional dysphagia therapy.
  Interventions: Other: Traditional Therapy

INTERVENTIONS:
Device: VitalStim — One group of children (Group A) will receive 24 sessions of NMES for combined with traditional therapy including oral motor exercises and laryngeal exercises will be performed to the participants. The equipment to be used for NMES is VitalStim®. VitalStim is a product of Empi®.
  Arms: VitalStim
Other: Traditional Therapy — The other group (Group B) will be receiving 24 sessions of traditional dysphagia therapy.
  Arms: Traditional therapy

SUMMARY:
Tracheostomy tubes are known to have a negative impact on swallowing. Dysphagia treatment includes using laryngoneuromuscular electrical muscular stimulation (LNMES). Evidence exist on the efficacy of LNMES in the treatment of dysphagia in adults, and scarce in pediatrics. There is no literature available for the efficacy of LNMES in the treatment of dysphagia on patients with tracheostomy tubes. The purpose of this study to determine the outcomes on dysphagia on children with tracheostomy tubes when treated using LNMES. Furthermore, the investigators aim to determine the relationship between parental stress and a child's modified diet.

ELIGIBILITY:
Inclusion Criteria:

PATIENT COHORT

* Children between 0-4 years 11 months
* Currently have tracheostomy tubes
* MBSS must indicate penetrations of more than 50% of swallows or aspiration of thin, ½ nectar-thick, nectar-thick or honey-thick liquids.
* The child must be on a modified diet of honey-thick liquids, nectar-thick liquids, ½ nectar-thick liquids, or no liquids by mouth.
* Able to tolerate a voice valve PARENT COHORT
* At least one primary caregiver of a qualifying child (see Child cohort).
* Parent/caregiver must be at least 18 years of age or older, provide primary care, and have medical decision making rights for the child.

Exclusion Criteria:

PATIENT COHORT

* Children who are not on modified diets or using a g-tube as an alternate means of nutrition
* Children with suspected or diagnosed heart problems
* Children with suspected or diagnosed epilepsy
* Children with a tendency to hemorrhage following acute trauma or fracture
* Children who have undergone recent surgical procedures when muscle contraction may disrupt the healing process
* Children for whom the LNMES would be: 1) over carotid sinus, 2) over neoplasm, 3) over active infection and 4) over areas of skin which lack normal sensation
* Children with difficulty tolerating tactile stimulation and tolerate the whole duration of the LNMES sessions.
* Children with difficulty tolerating tactile sensory stimulation such as tape and electrodes on the anterior aspect of the neck.

PARENT COHORT

* The caregiver that does not provide the primary care of the child and does not have medical decision making right
* Parents under 18

Ages: 30 Days to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-05-01 (Estimated); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
Assess Quality of Swallow during the MBSS (Modified Barium Swallow Study) using the Pen-Asp scale. | 3 months. LNMES intervention will be provided for 24 sessions during this time.
  The investigators will measure the change based on the patient's score of the Pen-Asp scale before and after the intervention provided.
Assess safety and adequate functional oral intake using the FOIS (Functional Oral Intake Scale) | 3 months. LNMES intervention will be provided for 24 sessions during this time.
  The investigators will measure the change based on the patient's score of the FOIS before and after the intervention provided.

SECONDARY OUTCOMES:
Assess Change in Parental Stress Level using the PSI-4 (Parent Stress Index-4) | 3 months
  Assess changes in parental stress level after treatments have been completed using the PSI-4 scale.

CONTACTS AND LOCATIONS:
Overall Officials: Aviril Sepulveda, Principal Investigator — Children's Hospital Los Angeles

IPD SHARING:
Plan to Share IPD: Undecided